CLINICAL TRIAL: NCT04369131
Title: Effect of Electrode Placement on Controlling Orthostatic Hypotension in People with Cervical Spinal Cord Injury
Brief Title: Controlling Orthostatic Hypotension in People with Cervical Spinal Cord Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled because none met the criteria.
Sponsor: Quality Living, Inc. (Other)
Responsible Party: Principal Investigator, Karen Hux, Ph.D., Director of Research, Quality Living, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Xcite study
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-01

CONDITIONS: Spinal Cord Injury Cervical; Hypotension, Orthostatic
Keywords: Spinal cord injury; Orthostatic hypotension; Functional electrical stimulation
MeSH Terms: conditions — Hypotension, Orthostatic; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Participants will engage in three baseline sessions to document blood pressure fluctuations associated with central nervous system dysregulation when changing from a sitting or supine position to a standing position involving the use of a head-up tilt table and no FES. Then, participants will engage in tilt table sessions in which the researchers randomly alternate the placement of FES pads across four conditions: (a) no FES, (b) calves only FES, (c) quads and abdominal only FES, and (d) calves, quads, and abdominal FES. Sessions will occur three to four times weekly until a participant demonstrates no OH upon tilt table adjustment to 90° (i.e., upright position) or the participant discharges from Quality Living, Inc., whichever comes first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): All participants will receive intervention in four conditions: (a) no FES, (b) calves only FES, (c) quads and abdominals only FES, and (d) calves, quads, and abdominals FES. Session-by-session alternation among conditions will occur in a unique, predetermined, randomized order for each participant.
  Interventions: Device: Functional electrical stimulation

INTERVENTIONS:
Device: Functional electrical stimulation — Randomized placement of FES pads in one of four locations during each session. Locations include: (a) none, (b) calves only, (c) quads and abdominals only, and (d) calves, quads, and abdominals.

SUMMARY:
A common therapeutic intervention after spinal cord injury (SCI) is prolonged standing in a standing frame. For people with SCI, standing for 40 minutes or more, three to four times weekly improves several health-related issues including well-being, circulation, skin integrity, reflex activity, bowel and bladder function, digestion, sleep, pain, and fatigue. However, a person who experiences orthostatic hypotension (OH)-defined as a decrease of 20mm hg in systolic blood pressure or a decrease of 10mm hg in diastolic pressure within 3 minutes of standing from a sitting or supine position-secondary to SCI may not tolerate positioning in a standing frame, thus resulting in a loss of access to these health benefits.

OH is common for people with SCI. It results from central nervous system dysregulation causing pooling of blood in the lower extremities that can lead to dizziness, light-headedness, blurred vision, weakness, fatigue, nausea, palpitations, headache, and/or syncope. Although an array of physical and pharmacologic interventions are available to people in the general population for managing OH, few such interventions have been evaluated for use by people with SCI, especially when the level of injury is C5 or above.

One possible intervention that may be effective for people with OH secondary to SCI is functional electrical stimulation (FES) because its application results in a dose-dependent increase in blood pressure. An unanswered question is whether the placement of FES electrodes on various parts of the body has differential effects. Therefore, the purpose of this study is to evaluate blood pressure responses among people with OH secondary to cervical SCI when receiving FES intervention involving the placement of electrodes in three different positions as well as when receiving no FES intervention during tilt table sessions. The selected positions for electrode placement are: (a) the calves, (b) the quads and abdominals, and (c) the quads, abdominals, and calves. The researchers hypothesize that FES intervention, regardless of placement, will result in better control of OH than no FES intervention and that no significant blood pressure difference will occur across the three FES placements.

DETAILED DESCRIPTION:
Participants will engage in three initial heads-up tilt table sessions with no FES intervention to confirm the presence and consistency of OH. During these sessions, the participant will lie supine on a tilt table at 0°, and, using a blood pressure cuff secured around the arm, the researchers will measure and record supine blood pressure. The researchers will then adjust the tilt table to 30° for three minutes and take and record another blood pressure measurement. If the participant reports no OH symptoms and the researchers observe no changes in appearance or signs of distress at that time, the researchers will query the participant about willingness to adjust the table to an additional 10° of tilt. Following three minutes at this level, the researchers will again measure and record the participant's blood pressure. These procedures will continue with increments of 10° of increased tilt every three minutes to a maximum of 90° tilt until the session time (maximum of 60 minutes) has elapsed or the participant expresses discomfort, measured blood pressure drops relative to the supine recording, or the researchers observe behaviors indicative of OH (e.g., sweating, change in skin color, change in breathing pattern, grimacing). If any of these OH symptoms occur, the researchers will adjust the tilt table to lower levels of incline until the participant's blood pressure stabilizes to the supine position measurement, and the session will be terminated.

Intervention sessions will begin after three days of baseline measurements. Intervention sessions will follow the same procedures except that the conditions will alternate randomly among the three FES placement and the no FES conditions. All sessions will be held at Quality Living, Inc., in Omaha, Nebraska.

ELIGIBILITY:
Inclusion Criteria:

* adult resident of Quality Living, Inc.
* SCI at the level of C5 or higher
* experience OH upon rising from a sitting or supine position
* comprehend English sufficiently to understand the consent form as measured by responses to included questions

Exclusion Criteria:

* any person who has a legally authorized representative responsible for making healthcare decisions because of compromised cognitive or communication status
* any person for whom FES is contraindicated as determined by the physiatrist responsible for monitoring the health and rehabilitation programs of Quality Living residents

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Change in tilt table angle from 0 degrees to maximum tolerated during session | Measured over the course of each one hour tilt table session
  Maximum tilt table angle, ranging from 0 to 90 degrees, tolerated by participant during each session
Change in blood pressure from initial reading at start of each tilt table session | Measured every three minutes throughout the time a participant is positioned on the tilt table
  Systolic and diastolic blood pressure values measured in millimeters of mercury

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hux, Ph.D., Principal Investigator — Quality Living, Inc.
Locations (1):
- Quality Living, Inc., Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chi L, Masani K, Miyatani M, Adam Thrasher T, Wayne Johnston K, Mardimae A, Kessler C, Fisher JA, Popovic MR. Cardiovascular response to functional electrical stimulation and dynamic tilt table therapy to improve orthostatic tolerance. J Electromyogr Kinesiol. 2008 Dec;18(6):900-7. doi: 10.1016/j.jelekin.2008.08.007. Epub 2008 Oct 2. PMID 18835189
- [Background] Eng JJ, Levins SM, Townson AF, Mah-Jones D, Bremner J, Huston G. Use of prolonged standing for individuals with spinal cord injuries. Phys Ther. 2001 Aug;81(8):1392-9. doi: 10.1093/ptj/81.8.1392. PMID 11509069
- [Background] Sampson EE, Burnham RS, Andrews BJ. Functional electrical stimulation effect on orthostatic hypotension after spinal cord injury. Arch Phys Med Rehabil. 2000 Feb;81(2):139-43. doi: 10.1016/s0003-9993(00)90131-x. PMID 10668765
- See also: Evaluation and Management of Orthostatic Hypotension — https://www.aafp.org/afp/2011/0901/p527.html